CLINICAL TRIAL: NCT05846659
Title: Phase 2 Randomized Clinical Trial Comparing the Safety and Efficacy of PULSAR-Integrated Radiotherapy + Pembrolizumab or Nivolumab Administered with or Without STING-Agonist IMSA101 in Patients with Oligoprogressive Solid Tumor Malignancies
Brief Title: Study of PULSAR-ICI +/- IMSA101 in Patients with Oligoprogressive Solid Tumor Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in ImmuneSensor corporate strategy
Sponsor: ImmuneSensor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMSA101-103
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Oligoprogressive
Keywords: Oligoprogressive solid tumor malignancies; Adult
MeSH Terms: interventions — Immune Checkpoint Inhibitors; pembrolizumab; Nivolumab; DEAE-Dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): PULSAR-ICI + IMSA101
  Interventions: Drug: IMSA101; Drug: Immune checkpoint inhibitor; Radiation: PULSAR
- Control Arm (Active Comparator): PULSAR-ICI
  Interventions: Drug: Immune checkpoint inhibitor; Radiation: PULSAR

INTERVENTIONS:
Drug: IMSA101 — Intra-tumoral administration once weekly for the first three weeks of Cycle 1 (Days 1, 8 and 15) and then on Day 1 of Cycles 2 and 3.
  Arms: Experimental Arm
Drug: Immune checkpoint inhibitor — 1st infusion on Cycle 1 Day 2, and then thereafter as per product label.
  Other Names: pembrolizumab; nivolumab
Radiation: PULSAR — 1st day of Cycles 1, 2 and 3.

SUMMARY:
Phase 2, open-label, multicenter, randomized study comparing the safety and efficacy of personalized ultra-fractionated stereotactic adaptive radiotherapy (PULSAR) combined with immune checkpoint inhibitor (ICI) immunotherapy (PULSAR-ICI) + IMSA101 and PULSAR-ICI alone in patients with oligoprogressive solid tumor malignancies after prior anti-cancer therapy.

DETAILED DESCRIPTION:
Patients shall be enrolled in 2 treatment arms as follows:

1. 15 patients in the control arm (PULSAR-ICI alone)
2. 30 patients in the experimental arm (PULSAR-ICI + IMSA101)

PULSAR-ICI with or without IMSA101 treatment will be administered to the patients in Cycles 1, 2, and 3, and thereafter only standard of care ICI monotherapy will be administered to all patients. Each treatment cycle will be 28 days in duration for Cycles 1, 2 and 3, then per standard of care monotherapy thereafter based on the product labels of the prescribed ICI.

The study will start with a safety run-in portion at 2 dose levels for the experimental arm, followed by a randomized portion for both treatment arms. The safety run-in shall employ a 3+3 safety run-in component.

All patients will be followed throughout the study for drug tolerability and safety by collecting clinical and laboratory data, including adverse events (AEs) using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 criteria, SAEs, concomitant medications, and vital signs.

All patients will be assessed for anti-tumor efficacy at screening, prior to the end of Cycle 3, and at 8-week intervals thereafter based on radiographic assessments (all outcome measures per RECIST Version 1.1 and iRECIST).

Tumor types and the corresponding treatment combinations to be evaluated will be identified prior to the first patient enrolled.

All patients will continue to receive their assigned treatment throughout the study until the occurrence of disease progression (based on iRECIST), death, or other unacceptable treatment-related toxicity, or until the study is closed by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Signed informed consent and mental capability to understand the informed consent
3. Histologically or cytologically documented solid tumor malignancies demonstrating new progression through prior anti-cancer therapy, with a prior 2 months of clinical stability (with at least Stable Disease), with radiographically documented presence of ≤ 6 metastatic lesions consistent with the diagnosis of "oligoprogressive" disease that are technically amenable to PULSAR
4. Patient's disease must be evaluable per RECIST Version 1.1
5. All metastatic lesions amenable to administration of radiotherapy, at the discretion of the investigator
6. Must have at least one single pre-defined progressing lesion/lesion site (longest diameter ≥ 10 mm and ≤ 50 mm) suitable for intra-tumoral injection
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
8. Electrocardiogram (ECG) without evidence of clinically meaningful conduction abnormalities or active ischemia as determined by the investigator
9. Acceptable organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) > 1,500 cells/μL
   * Platelets > 50,000 cells/μL
   * Total bilirubin ≤ 1.5 times (×) the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransaminase (ALT) ≤ 2.5 × ULN. If liver metastases are present, AST/ALT < 5 × ULN
   * Serum creatinine < 1.5 mg/dL and a measured creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault formula
   * Prothrombin time (PT)/partial thromboplastin time (PTT) ≤ 1.5 × ULN
10. Women of child-bearing potential (defined as a female who has experienced menarche and who has not undergone successful surgical sterilization [hysterectomy, bilateral salpingectomy, or bilateral oophorectomy]) or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months with an appropriate clinical profile at the appropriate age, eg, greater than 45 years) must have a negative serum pregnancy test prior to first dose of study treatment
11. Male and female patients with reproductive potential must agree to use two forms of highly effective contraception throughout the study

Exclusion Criteria:

1. Prior receipt of stimulator of interferon genes (STING) agonist
2. Prior receipt of therapeutic radiotherapy to all progressive lesions intended for PULSAR treatment
3. Anti-cancer therapy, except pembrolizumab and nivolumab, within 4 weeks or < 5 half-lives of the first dose of study treatment
4. Existence of primary tumor that requires therapeutic treatment beyond the provided immune checkpoint inhibitor drug
5. Failure to recover, to Grade 1 or less, from clinically significant AEs due to prior anti-cancer therapy, as judged by the investigator
6. Previous life-threatening (Grade 4) immune-related adverse event (irAE)
7. Known untreated brain metastases or treated brain metastases that have not been stable (scan showing no worsening of central nervous system [CNS] lesion[s] and no requirement of corticosteroids) ≥ 4 weeks prior to study enrollment
8. Existence of actionable mutations that are eligible for a mutation-targeting drug that represents standard-of-care
9. Baseline prolongation of QT/corrected QT (QTc) interval (QTc interval > 470)
10. Uncontrolled intercurrent illness (including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations) that in the opinion of the investigator would limit compliance with study requirements
11. Women who are pregnant or breastfeeding
12. Sponsor reserves the right to exclude any patient from the study on the basis of pre-study medical histories, physical examination findings, clinical laboratory results, prior medications, or other entrance criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Anti-tumor effects | assessment at 12 months
  Progression-free rate at 12 months

SECONDARY OUTCOMES:
Safety and tolerability | upon enrolment through end of study period (2 years)
  Occurrence of treatment-related adverse events and SAEs
Anti-tumor effects | 6 to 22 months
  Progression-free at 8-week intervals from 6 months to 22 months
Anti-tumor effects | upon enrolment through end of study period (2 years)
  Time-to-progression (TTP)
Anti-tumor effects | upon enrolment through end of study period (2 years)
  Overall response rate, duration of response, progression-free survival
Quality of life (QoL) | upon enrolment through end of study period (2 years)
  Patient-reported outcome using FACT-G

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Widhelm, Study Director — ImmuneSensor Therapeutics
Locations (14):
- United States (14):
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital/Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No